CLINICAL TRIAL: NCT03955016
Title: A Randomized Controlled Trial to Evaluate the Effect of a Rehabilitation Program on the Exercise Capacity of Patients With Pulmonary Hypertension
Brief Title: Rehabilitation for Patients With Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Wim Janssens, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S61141
Record Dates: First submitted 2018-07-16; First posted 2019-05-17 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary rehabilitation; physical activity
MeSH Terms: conditions — Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded for the outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): 15 weeks pulmonary rehabilitation program consisting of 2 weeks inpatient, 2 weeks outpatient and 11 weeks home-based rehabilitation.
  Interventions: Other: Pulmonary rehabilitation
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Pulmonary rehabilitation — Rehabilitation program consisting of 2 weeks inpatient (supervised training 5 times per week), 2 weeks outpatient (supervised sessions 3 times per week) and 11 weeks home-based exercise training (weekly phone call).
  During the inpatient phase, patients will receive on top of the supervised training sessions a consultation of the dietitian, PH psychologist, social worker and specialized nurse. During the ambulatory rehabilitation phase patients will have 2 session with the occupational therapist.
  Every supervised training session contains:
  1. Interval training on a cyclo-ergometer
  2. Strength training of the upper and lower extremities
  3. Guided walks
  Arms: Rehabilitation group

SUMMARY:
The purpose of this study is to test the impact of a personalized, partly supervised rehabilitation program on the exercise capacity in patients with pulmonary hypertension. The rehabilitation program consists of 2 weeks inpatient, 2 weeks ambulatory and 11 weeks home based rehabilitation.

DETAILED DESCRIPTION:
The present study is a 15 weeks, randomized (1:1) controlled trial. Patients in both groups will not change their usual medical treatment. After 2 clinical visits (screening and randomization visit), patients in the intervention group will follow a 15 week rehabilitation program consisting of 2 weeks inpatient, 2 weeks outpatient and 11 weeks home based rehabilitation. At the end of the outpatient rehabilitation phase (week 4) and the home-based program (week 15), clinical outcomes will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years
* Pulmonary arterial hypertension (PAH, Group 1 of Nice classification) and chronic thromboembolic pulmonary hypertension (CTEPH, group 4)
* WHO functional class II-III
* PH diagnosed by right heart catheter showing:

  1. Baseline mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
  2. Baseline pulmonary vascular resistance (PVR) ≥ 240dyn x s x cm-5
  3. Baseline pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHgg
* Patients receiving optimized conventional PH therapy including intensified treatment with diuretics and who have been stable for 2 months before entering the study.
* Except for diuretics, medical treatment should not be expected to change during the entire 15-week study period.
* Negative pregnancy test (β-HCG) at the start of the trial and appropriate contraception throughout the study for women with child- bearing potential
* Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria:

* PH of any cause other than permitted in the entry criteria, e.g. concomitantly to portal hypertension, complex congenital heart disease, reversed shunt, HIV infection, suspected pulmonary veno-occlusive disease based on pulmonary edema during a previous vasoreactivity test or on abnormal findings compatible with this diagnosis (septal lines or pulmonary edema at high resolution computer tomography), congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension or unclear diagnosis
* Patients with signs of right heart decompensation
* Walking disability
* Acute infection, pyrexia
* Any change in disease-targeted therapy within the last 2 months
* Any subject who is scheduled to receive an investigational drug during the course of this study
* Severe lung disease: FEV1/FVC <0.5 and total lung capacity <70% of the normal value
* Active myocarditis, instable angina pectoris, exercise induced ventricular arrhythmias, decompensated heart failure, active liver disease, porphyria or elevations of serum transaminases >3 x ULN (upper limit of normal) or bilirubin >1.5 x ULN
* Hemoglobin concentration of less than 75% of the lower limit of normal
* Systolic blood pressure <85 mmHg
* History or suspicion of inability to cooperate adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional exercise capacity | Baseline, 4 weeks, 15 weeks
  Change in six minutes-walk distance measured at baseline, after 4 weeks and at the end of the study (15 weeks after randomization).

SECONDARY OUTCOMES:
Difference in change over time between the rehabilitation and the control group in SF-36 | Baseline, 4 weeks, 15 weeks
  Health related quality of life (HRQoL) will be measured by the extensively validated generic HRQoL questionnaire, the 36-Item Short Form Survey Instrument (SF-36). This questionnaire includes two main scores with a physical component and an emotional component scale and eight subscales. The score ranges between 0 and 100, higher scores indicate a better quality of life. The questionnaire is self-administered and will be completed on paper
Difference in change over time between the rehabilitation and the control group in EmPHasis-10. | Baseline, 4 weeks, 15 weeks
  Health related quality of life (HRQoL) will be measured the EmPHasis-10 questionnaire, measuring the impact of PH on health related quality of life. The score ranges between 0 and 50, higher scores indicate worse quality of life.
Change from baseline to 15 weeks between the rehabilitation and the control group in WHO functional class | Baseline, 15 weeks
  The WHO functional classification ranges from class I (patients with PH but without resting limitation of physical activity) to class IV (patients with PH with inability to carry out any physical activity without symptoms). The WHO functional class is a powerful predictor of survival in patients with PH.
Difference in change over time between the rehabilitation and the control group in Borgscale at the end of the 6MWD test | Baseline, 4 weeks, 15 weeks
  Borg (0-10) scale reporting on dyspnea and fatigue will be administered at the end of the six-minutes walk test. The score ranges between 0 and 10, a higher score means more symptoms of dyspnea / fatigue.
Change from baseline to 15 weeks between the rehabilitation and the control group in maximal exercise capacity | Baseline, 15 weeks
  Maximal exercise capacity will be assessed by a maximal incremental cycling test. After a 2-min resting period and 3 minutes of unloaded cycling, the patients will start at 20 W and cycle until symptom limitation at an incremental workload of 10 W/min. Oxygen consumption, carbon dioxide output and ventilation will be measured breath by breath (Vmax series, SensorMedics, Anaheim, CA). Heart rate and oxygen saturation will be registered continuously. Peak workload, oxygen consumption (VO2 max), heart rate, blood pressure, oxygen saturation, ventilation and VE/VCO2 slope will be retrieved.
Difference in change over time between the rehabilitation and the control group in Objectively measured physical activity | Baseline, 4 weeks, 15 weeks
  At every time point, physical activity will be measured for 1 week, using a physical activity monitor validated to be used in patients with respiratory disease. Patients will be asked to wear the monitor during waking hours. The mean number of steps per day and time spent in activities of at least moderate intensity will be retrieved as outcomes.
Difference in change over time between the rehabilitation and the control group in symptoms of anxiety and depression (HADs questionnaire) | Baseline, 4 weeks, 15 weeks
  Symptoms of anxiety and depression will be assessed by the Depression, Anxiety, and Stress Scale. This questionnaires is self-administered and will be completed on paper. Higher scores indicate more symptoms of anxiety / depression.
Difference in change over time between the rehabilitation and the control group in Isometric quadriceps force | Baseline, 4 wekes, 15 weeks
  An isometric maximal volitional contraction of the right quadriceps muscle be performed using the Biodex dynamometer with the patient seated with a 90° hip and 60° knee flexion. The best of 3 reproducible measurements will be retrieved as a measure of quadriceps force.
Change from baseline to 15 weeks between the rehabilitation and the control group in hemodynamics measured by echocardiography | Baseline, 15 weeks
  Hemodynamics measured by echocardiography at rest and during a symptom limiting exercise test. The following outcomes will be investigated: Change in tricuspid annular plane systolic excursion, Change in tissue Doppler imaging, Change in left ventricular pump function, Change in right ventricular pump function , Change in thickness of interventricular septum, Change insize of inferior vena cava, Change in systolic pulmonary arterial pressure, Change in left ventricular eccentricity index, Change in Tei index , Change in right ventricular area, Change in right atrial area
Change from baseline to 15 weeks between the rehabilitation and the control group in proportion of patients who exceeded the MID in 6MWD | Baseline, 15 weeks
  MID will be defined as an increase of at least 30m
Change from baseline to 15 weeks between the rehabilitation and the control group in heart function as measured by MRI (optional) | Baseline, 15 weeks
  MRI scan at rest and during exercise combined with right heart catherization and blood sampling before and after the exercise protocol.
adverse events | 15 weeks
  Patients will be asked about visits to general practitioner and hospitalizations due to any medical reasons in order to control the occurrence of adverse events. In a semi-structured way,, occurrence of exercise related and non-exercise related adverse events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof, Principal Investigator — University hospitals Leuven, KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided